CLINICAL TRIAL: NCT04342312
Title: Intensive Molecular and Electropathological Characterization of patientS undergOing atriaL fibrillATion ablatION: a Multicenter Prospective Cohort Study
Brief Title: Intensive Molecular and Electropathological Characterization of Patients Undergoing Atrial Fibrillation Ablation
Acronym: ISOLATION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University (Other)
Collaborators: Maastricht University Medical Center (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL70787.068.19
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation Paroxysmal; Atrial Fibrillation, Persistent
Keywords: Pulmonary Vein Isolation; Cryoballoon ablation; Radiofrequency ablation; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pulmonary vein isolation — Participation in this study does not influence the choice of ablation technique. Usually, cryoballoon ablation is chosen for patients with paroxysmal AF and no previous ablations. Radiofrequency ablation is often used for redo procedures or for patients with persistent AF. Hybrid ablations are most applied in persistent AF patients. However, physicians may deviate from these standard approaches for a variety of reasons, including personal experience or preference.
  Other Names: atrial fibrillation ablation; AF ablation

SUMMARY:
Rationale:

Although there are several individual factors which are known to influence the chances of successful atrial fibrillation (AF) ablation, it remains a challenge to identify patients at risk for ablation failure with satisfactory certainty.

Objectives:

To identify predictors of success of AF ablation including clinical factors, AF recurrence patterns, anatomical and electrophysiological characteristics, circulating biomarkers and individual genetic background.

Study design:

Prospective registry of patients undergoing AF ablation. Clinical characteristics and results of routine tests are collected. In addition, the following (non-standard) tests are performed: extended surface electrocardiogram (extECG), extended rhythm monitoring, biomarker testing, genetic analysis, questionnaires. In subgroups of patients transesophageal electrocardiogram (TE-ECG), epicardial electroanatomical mapping and/or left atrial appendage (LAA) biopsy is performed.

Study population:

Patients aged 18 years and older with documented AF, scheduled for AF ablation.

Main study endpoints:

Ablation success after 12 and 24 months, defined as freedom from any episode of documented atrial arrhythmia after the blanking period.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Documented atrial fibrillation;
* Scheduled for AF ablation or redo AF ablation;
* Able and willing to provide written informed consent.

Exclusion criteria

* Serious patient condition before ablation;
* Physically or mentally unable to provide written informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All eligible patients scheduled for AF ablation of at the MUMC+ and Radboudumc will be asked to participate in this cohort study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Ablation success | 12 months
  Ablation success is defined as freedom from documented recurrence of atrial arrhythmia after 12 months. Recurrences in the first 3 months after the index procedure (blanking period) are exempted.
  Atrial arrhythmias are AF, atrial tachycardia (AT) and non-isthmus dependent atrial flutter (AFl), lasting more than 30 seconds, documented on ECG or Holter monitoring.

SECONDARY OUTCOMES:
Time to recurrence of AF or atrial arrhythmia after the blanking period | 24 months
Early recurrences of AF or atrial arrhythmia, defined as any episode of AF AT or non-isthmus dependent AFl during the blanking period. | 3 months
Disease progression to persistent or permanent AF. | 24 months
Changes in circulating biomarkers and non-invasive electrophysiological markers for substrate quantification. | 12 months
Use of antiarrhythmic drugs (AADs) one year after ablation. | 12 months
Number of veins with pulmonary vein reconnection at redo procedure. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schotten, MD PhD, Study Chair — Maastricht University, departments of physiology and cardiology; Kevin Vernooy, MD PhD, Study Chair — Maastricht UMC+ and Radboudumc, department of cardiology
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - Maastricht UMC+, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Betz K, Verhaert DVM, Gawalko M, Hermans ANL, Habibi Z, Pluymaekers NAHA, van der Velden RMJ, Homberg M, Philippens S, Hereijgers MJM, Vorstermans B, Simons SO, den Uijl DW, Chaldoupi SM, Luermans JGLM, Westra SW, Lankveld T, van Steenwijk RP, Hol B, Schotten U, Vernooy K, Hendriks JM, Linz D. Atrial fibrillation-specific refinement of the STOP-Bang sleep apnoea screening questionnaire: insights from the Virtual-SAFARI study. Clin Res Cardiol. 2023 Jun;112(6):834-845. doi: 10.1007/s00392-023-02157-9. Epub 2023 Feb 11. PMID 36773038